CLINICAL TRIAL: NCT00330967
Title: Mechanisms of Insulin Resistance in Humans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: ENDA-029-05F
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Inflammation; Insulin Resistance
Keywords: Fat Emulsions, Intravenous; Free Fatty Acids; Glucose Clamp Technique; Inflammation; Insulin Resistance; Muscle, Skeletal; NF-Kappa B
MeSH Terms: conditions — Inflammation; Insulin Resistance | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples, muscle biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: healthy subjects
  Interventions: Drug: 20% Intralipid
- Group 2: healthy subjects different from group 1
  Interventions: Drug: 20% Intralipid

INTERVENTIONS:
Drug: 20% Intralipid — lipid infusion

SUMMARY:
The Objectives of the study are to: (1)compare the inflammatory response and insulin resistance in skeletal muscles during a systemic infusion of lipid with that during a local infusion of lipid into the femoral artery. which would cause minimal or no systemic hyperlipidemia but local plasma free fatty acid (FFA) concentrations similar to those during the systemic lipid infusion, and (2) determine the inflammatory response and insulin resistance in skeletal muscle during an infusion of lipid into the femoral artery as described above after NF-KB inhibition by high dose salicylate treatment in humans.

DETAILED DESCRIPTION:
Insulin resistance in skeletal muscle is a characteristic abnormality in obesity and the metabolic syndrome and a major factor responsible for the development of type 2 diabetes. Although the mechanisms responsible for muscle insulin resistance are largely unclear, lipid oversupply is an important factor. Among numerous potential mechanisms whereby lipid oversupply may cause muscle insulin resistance, current evidence points towards inflammation as being critical. Recent studies in animals, however, indicate that the inflammatory response in skeletal muscles may require the presence of circulating pro-inflammatory factors suggesting that the inflammation induced insulin resistance in skeletal muscles may be a secondary event. More specifically, activation of Nuclear Factor-Kappa B(NF-kB), and inflammatory master switch that drives the production of numerous pro-inflammatory cytokines in fat and liver, has been implicated in causing insulin resistance in skeletal muscles by increasing circulating pro-inflammatory cytokines. In contrast, animal studies have found that activation of NF-KB directly in skeletal muscles has no or little effect on its insulin sensitivity but does produce other abnormalities such as increased proteasome activity. The study shall therefore be undertaken to determine to what extent lipid-induced inflammation and insulin resistance in skeletal muscles requires the presence of circulating proinflammatory factors in humans.

ELIGIBILITY:
Inclusion Criteria:

* two groups of 16 healthy subjects

Exclusion Criteria:

* diabetes or impaired glucose tolerance
* peripheral vascular disease
* pulmonary disease
* clinically significant hepatic or renal disease
* triglycerides >200mg/dl
* anemia
* abnormal PT, PTT or INR
* pregnancy or lactation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-04; Primary Completion 2012-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Oh, MD, Principal Investigator — Phoenix VA Health Care System Carl T. Hayden VA Medical Center, Phoenix, AZ
Locations (1):
- Phoenix VA Health Care System Carl T. Hayden VA Medical Center, Phoenix, AZ, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Systemic Intralipid infusion subjects
  20% Intralipid: lipid infusion
- Group 2: Femoral arterial Intralipid infusion subjects
  20% Intralipid: lipid infusion
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 0 | 25
Completed | 0 | 11
Not Completed | 0 | 14
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Physician Decision | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Femoral Intralipid infusion subjects
  20% Intralipid: lipid infusion
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 0 | 25 | 25
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 25 | 25
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 47.65 (11.43) | 47.65 (11.43)
Gender [Number; unit: participants]
  Female |  | 4 | 4
  Male |  | 21 | 21
Region of Enrollment [Number; unit: participants]
  United States |  | 25 | 25

OUTCOME MEASURES:

1. Primary Outcome: Insulin Signaling With Lipid Infusion
Description: IRS-1 expression in response to femoral lipid infusion in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blot bands, normalized to a housekeeping protein, GAPDH, in control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  IRS-1 Basal | 0.4334 (0.2199)
  IRS-1 Basal Lipid | 0.7276 (0.0173)
  IRS-1 Insulin | 0.5264 (0.3810)
  IRS-1 Insulin Lipid | 0.3534 (0.1391)

2. Primary Outcome: Phos-p38 MAPK Expression With Femoral Lipid and Insulin Infusions
Description: Phosphorylation of p38 MAPK in response to femoral lipid and insulin infusions. phospho-p38 MAPK expression in response to femoral lipid infusion in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blots, normalized to a housekeeping protein, GAPDH, of control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Group 2: Femoral Intralipid infusion group
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  Phos-p38 MAPK Basal | 0.000394 (0.000164)
  Phos-p38 MAPK Basal Lipid | 0.001271 (0.001013)
  Phos-p38 MAPK Insulin | 0.000337 (0.000140)
  Phos-p38 MAPK Insulin Lipid | 0.000270 (0.000049)

3. Primary Outcome: p38 MAPK Expression With Femoral Lipid and Insulin Infusions
Description: p38 MAPK expression in response to femoral lipid and insulin infusions in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blots, normalized to a housekeeping protein, GAPDH, of control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  p38 MAPK Basal | 0.000455 (0.0000088)
  p38 MAPK Basal Lipid | 0.001291 (0.0008)
  p38 MAPK Insulin | 0.000502 (0.000337)
  p38 MAPK Insulin Lipid | 0.000377 (0.0000903)

4. Primary Outcome: Phospho-ERK MAPK Expression With Femoral Lipid and Insulin Infusions
Description: Phosphorylation of ERK MAPK in response to femoral lipid and insulin infusions in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blots, normalized to a housekeeping protein, GAPDH, of control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  Phos-ERK MAPK Basal | 0.000091 (0.0000378)
  Phos-ERK MAPK Basal Lipid | 0.000108 (0.0000366)
  Phos-ERK MAPK Insulin | 0.000096 (0.0000103)
  Phos-ERK MAPK Insulin Lipid | 0.000092 (0.0000070)

5. Primary Outcome: ERK MAPK Expression With Femoral Lipid and Insulin Infusions
Description: ERK MAPK expression in response to femoral lipid and insulin infusions in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blots, normalized to a housekeeping protein, GAPDH, of control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  ERK MAPK Basal | 0.000103 (0.0000722)
  ERK MAPK Basal Lipid | 0.000158 (0.0000826)
  ERK MAPK Insulin | 0.000124 (0.0000237)
  ERK MAPK Insulin Lipid | 0.000114 (0.0000017)

6. Primary Outcome: Phospho-JNK MAPK Expression With Femoral Lipid and Insulin Infusions
Description: Phosphorylation of JNK MAPK in response to femoral lipid and insulin infusions in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blots, normalized to a housekeeping protein, GAPDH, of control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  Phos-JNK MAPK Basal | 0.00401 (0.002967)
  Phos-JNK MAPK Basal Lipid | 0.005888 (0.004952)
  Phos-JNK MAPK Insulin | 0.003756 (0.002537)
  Phos-JNK MAPK Insulin Lipid | 0.00224 (0.001161)

7. Primary Outcome: JNK MAPK Expression With Femoral Lipid and Insulin Infusions
Description: JNK MAPK expression in response to femoral lipid and insulin infusions in skeletal muscle. Relative protein expression was calculated by densitometry analysis of Western blots, normalized to a housekeeping protein, GAPDH, of control and treated groups.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2
Number analyzed (Participants) | 2
ratio
  JNK MAPK Basal | 0.001364 (0.00594)
  JNK MAPK Basal Lipid | 0.002996 (0.002837)
  JNK MAPK Insulin | 0.002151 (0.002032)
  JNK MAPK Insulin Lipid | 0.001783 (0.001883)

ADVERSE EVENTS:
Groups:
- Group 1: Systemic Intralipid infusion group
  20% Intralipid: lipid infusion
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/25
Other Adverse Events (participants affected / at risk) | 0/0 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=0) | Group 2 (N=25)
Edema (Surgical and medical procedures) | 0 (0) | 1 (1) — Right lower extremity edema following muscle biopsy.

LIMITATIONS AND CAVEATS:
The study's original Principal Investigator left the VA prior to the completion of data acquisition and no further subjects were enrolled. The data entered were analyzed based solely on study files in the system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No